CLINICAL TRIAL: NCT03915314
Title: The Association Between Blood Biomarkers and Postoperative Delirium in Elective Non-Cardiac Surgery Under General Anesthsia.
Brief Title: Correlation Between Blood Biomarkers and Postoperative Delirium in Elective Non-Cardiac Surgery.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Han Yuan, Director, Xuzhou Medical University
Other Study IDs: XYFY2018-KL091-01
Record Dates: First submitted 2019-04-05; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Delirium; Elective Non-Cardiac Surgery
Keywords: delirium; blood biomakers; endothelial dysfunction; blood brain barrier (BBB)
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine and blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POD group: POD group refers to the patients who were diagnosed to be delirious by the Confusion Assessment Method.
  Interventions: Diagnostic Test: Neuropsychological tests
- Non-POD group: Non-POD refered to the patients who did not become delirious by the Confusion Assessment Method.
  Interventions: Diagnostic Test: Neuropsychological tests

INTERVENTIONS:
Diagnostic Test: Neuropsychological tests — The investigators do the neuropsychological tests, Mini-Mental score examination (MMSE),Charlson Comorbidity Index(CCI)，Quality of Recovery Score - 40 (QoR-40),CAGE Alcoholism Questionnaire,blood albumin、hemoglobin content、ALT、AST、BUN、Cr、1 day before the surgery（baseline);serum biomarkers of endothelial dysfunction，blood brain barrier disruption and neuronal injury to be measured at 2 time points,1 day before the surgery（baseline）and postoperative day 1； Confusion Assessment Method（CAM)，Numerical Rating Scale（NRS）once before discharge from PACU and 1、2、3 days after surgery twice a day； QoR-40 1 day after surgery.

SUMMARY:
More than 20% of patients over 60 years old develop postoperative delirium following non-cardiac surgery . Delirium increases morbidity and mortality , and may lead to long-term cognitive impairment . The underlying mechanisms behind delirium are not understood , endothelial dysfunction and disruption of the blood brain barrier (BBB ) caused by perioperative systemic inflammation may play a important role in the development of delirium . This study intends to evaluate the relationship between neuroinflammation and postoperative delirium in elderly non-cardiac surgery patients . The results of the study are to identify risk factors and explore the biomarkers most closely linked to each step of the proposed pathway .

DETAILED DESCRIPTION:
The investigators do the neuropsychological tests , Mini-Mental score examination (MMSE ) , Charlson Comorbidity Index (CCI ) , Quality of Recovery Score - 40 (QoR-40 ) 1 day before the surgery（baseline ) . Serum of the patients was collected before operation and at POD1 , and then detect the concentration change of biomarkers of endothelial dysfunction , blood brain barrier disruption and neuronal injury . Also , the patients were interviewed once before discharge from PACU and twice on postoperative days 1-3 by the Confusion Assessment Method and then divided them into POD and non-POD groups . Meanwhile , the severity of pain (Numerical Rating Scale（NRS )) was evaluated at the same time and QoR-40 at 1 day after surgery .

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing selective major noncardiac surgery and general anesthesia;
2. Age 60-90 yrs;
3. Anesthesia Society of American (ASA) Scale II~III;
4. Anticipated surgery time 2-6 hrs
5. Written informed consent;

Exclusion Criteria:

1. decline to participate
2. Dementia patients（Mini-mental state examination< 20）
3. Factors existed that affect cognition assessment such as language,visual,and auditory dysfunction.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥60 years undergoing elective non-cardiac major surgery under general anesthesia were investigated.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
serum concentration change in biomarker of endothelial dysfunction | baseline, postoperative day 1
  C-terminal endothelin-1 (CT-proET-1) to be measured at 2 time points
serum concentration change in biomarker of blood brain barrier disruption | baseline, postoperative day 1
  caveolin-1 to be measured at 2 time points
serum concentration change in biomarker of neuronal injury | baseline, postoperative day 1
  Neurofilament light (NfL) to be measured at 2 time points
The incidence of postoperative delirium | From day 0 to up to 3 days after the surgery
  The patients were interviewed one day before the surgery and on postoperative days 1-3 by the Confusion Assessment Method and then divided them into POD and non-POD groups.

SECONDARY OUTCOMES:
Quality of Recovery Score - 40 (QoR-40) at baseline | 1 day before the surgery(baseline)
  Quality of recovery will be evaluated by Quality of Recovery 40 (QoR40),which assesses five dimensions of recovery (physical comfort,emotional state, physical independence , physiological support and pain ). Each item is rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).
Quality of Recovery Score - 40 (QoR-40) after surgry | 1 day after the surgery
  Quality of recovery will be evaluated by Quality of Recovery 40 (QoR40),which assesses five dimensions of recovery (physical comfort,emotional state, physical independence , physiological support and pain ). Each item is rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).
The severity of pain at baseline | 1 day before the surgery(baseline)
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.
The severity of pain after surgry | From day 0 to up to 3 days after the surgery
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Junli Cao, Xuzhou, Jiangsu, China